CLINICAL TRIAL: NCT05346822
Title: The Effects of a Patient-specific Integrated Education Program on Pain, Perioperative Anxiety, and Functional Recovery Following Total Knee Replacement
Brief Title: The Efficacy of Collaborative Patient Education on Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KMUHIRB-E(I)-20190255
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Knee Arthritis
Keywords: integrated rehabilitation; total knee arthroplasty; personalized medicine

STUDY DESIGN:
Intervention Model Description: A two-site, two-arm, parallel-group controlled trial of integrated rehabilitation program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- integrated rehabilitation program for total knee arthroplasty (Experimental): the intervention was performed in one KMUH affiliated facility
  Interventions: Procedure: integrated rehabilitation (the collaborative patient education)
- normal total knee arthroplasty clinical pathway (No Intervention): no integrated rehabilitatoin program for total knee arthroplasty patients with our conventional clinical pathway

INTERVENTIONS:
Procedure: integrated rehabilitation (the collaborative patient education) — Pre-operative education and rehabilitation. During hospitalization: group rehabilitation education program. Discharge: post-operative care navigation for total knee arthroplasty
  Arms: integrated rehabilitation program for total knee arthroplasty

SUMMARY:
This project is about the integrated rehabilitation program for the patients receiving total knee arthroplasty. The investigators are monitoring the WOMAC(Western Ontario and Mcmaster University Arthritis Index)/ Pain scores/Anxiety scores/Knee society scores in the treatment course between the intervention group and the control group.

DETAILED DESCRIPTION:
This is a quasi-experimental design study. The participants received total knee arthroplasty by one single surgeon in two facilities within the same medical system (Kaohsiung Medical University affiliated hospitals). The intervention groups received integrated rehabilitation program including verbal one-on-one education, personalized post-operation rehabilitation during admission and scheduled post-operation follow up by a nurse case manager. The control group received the same surgery with traditional clinical pathway by the single surgeon in another affiliated hospital.

We recorded the pain scores, state-trait anxiety inventory scores, WOMAC(Western Ontario and Mcmaster Universities Arthritis Index) scores, American Knee society scores for these participants.

ELIGIBILITY:
Inclusion Criteria

* Patients over 65 years of age
* Patients scheduled to receive unilateral total knee arthroplasty due to advanced osteoarthritis
* Patients are able to understand the study and express opinions clearly
* Patients are willing to participate in this study and provide informed consents

Exclusion Criteria

* Patients with inflammatory joint disease
* Patients with neurosensory system disease (such as stroke or parkinsonism)
* Patients have intellectual impairment, or dementia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Pain Score (VAS) | From admission to 3 months after surgery
  Minimum pain intensity from 0 to Maximum of 10. Higher scores mean a higher pain intensity.
State-trait Anxiety Inventory (STAI) | From admission to 3 months after surgery
  Peri-operative anxiety scoring system. STAI varies from a minimum score of 20 to a maximum score of 80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80). Higher scores mean higher anxiety.
American Knee Society Scores(AKS) | From admission to 3 months after surgery
  The AKS ranges from 100 (normal knee function score) to 0 (worst knee function score). Higher scores mean a better outcome.
WOMAC (Western Ontario and Mcmaster Universities Arthritis Index) | From admission to 3 months after surgery
  The WOMAC evaluates 3 dimensions : pain(maximal score of 20), stiffness(maximal score of 8), and physical function(maximal score of 68). Higher scores mean worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No sharing of the individual participant data